CLINICAL TRIAL: NCT07057596
Title: Neoadjuvant Tebentafusp in Patients With Metastatic Uveal Melanoma
Acronym: NEO-TB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español Multidisciplinar de Melanoma (Other)
Collaborators: INMUNOCORE (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEM 2302; 2023-509076-42-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Mestastatic Uveal Melanoma
Keywords: Melanoma; Tebentafusp; Metastatic; Neoadjuvant
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — tebentafusp

STUDY DESIGN:
Intervention Model Description: NEO-TB is a non-randomized, single arm, multi-centre, phase II study of Tebentafusp monotherapy in subjects with resectable / potentially resectable disease within the liver and absence of extra-liver disease.
  The trial will enroll 19 patient male and female, ≥ 18 years, with ECOG PS 0-1 patients with metastatic uveal melanoma (HLA)-A*02:01 positive who have resectable or potentially resectable metastatic lesions only in the liver.
  The study is divided into 4 phases: Screening, Treatment, Surgery and Follow-up. All patients will undergo periodic tumor assessments by Computed Tomography (TC) o Magnetic Resonance Imaging (MRI) scan every 8 weeks ± 7 days from the start of study treatment and during the first 48 weeks of study. Tumor assessments will be performed every 12 weeks ± 7 days thereafter until relapse or patient withdrawal. After surgery, CT or MRI scans will be performed every 12 weeks ± 7 days thereafter, regardless of time after study inclusion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Tebentafusp (Experimental): Patients will receive tebentafusp intravenously (IV) weekly for 6 months with liver directed imaging every 2 months to identify rapid progressors. Rapid progressors will discontinue tebentafusp and have surgical resection if considered feasible. After 6 months, patients with complete response (CR) according to RECIST will continue tebentafusp therapy. Surgery might be an option if deem appropriate by local PI); while patients achieving partial response or stable disease will be evaluated for tumor resection and will enter into Surgery phase. Surgery will be conducted 7 months (+/- 1 month). If progressioh disease (PD) occurs earlier surgery can happen earlier. After surgery, patients without pCR or R0 surgery will maintain tebentafusp until disease relapse, unacceptable toxicity or patient withdrawal. Patients with pCR and R0 will continue tebentafusp therapy for 1 additional year or until disease relapse, unacceptable toxicity or patient withdrawal.
  Interventions: Drug: Tebentafusp

INTERVENTIONS:
Drug: Tebentafusp — Patients will receive tebentafusp intravenously (IV) weekly for 6 months with liver directed imaging every 2 months to identify rapid progressors. Tebentafusp will be administered at 20 micrograms on W1D1, 30 micrograms on W2D1, and 68 micrograms once every week thereafter.
  After 6 months, patients with complete response (CR) according to RECIST will continue tebentafusp therapy (surgery might be an option if deem appropriate by local PI); while patients achieving partial response or stable disease will be evaluated for tumor resection and will enter into Surgery phase. Surgery will be conducted 7 months (+/- 1 month). If progressioh disease (PD) occurs earlier surgery can happen earlier. After surgery, patients without pCR or R0 surgery will maintain tebentafusp until disease relapse, unacceptable toxicity or patient withdrawal. Patients with pCR and R0 will continue tebentafusp therapy for 1 additional year or until disease relapse, unacceptable toxicity or patient withdrawal.

SUMMARY:
Uveal melanoma (UM) is a rare type of melanoma, with an incidence of 4.4 cases per million in Europe each year. During recent years, different treatment approaches have been tested in patients with metastatic UM. Responses have been reported primarily with localized treatment in patients with a limited number of liver metastases. In cases of diffuse liver involvement or extrahepatic disease, systemic therapies are justified. However, to date, systemic therapies such as targeted therapy with selumetinib or conventional chemotherapy have failed in metastatic UM.

Neo-TB is a Phase II, single arm, multicentre clinical trial designed to evaluate efficacy and safety of tebentafusp used as a single agent in patients with metastatic uveal melanoma with resectable / potentially resectable liver metastasis and absence of extrahepatic disease.

The main questions it aims to answer are:

1. Which is the capacity of tebentafusp used as a single agent to generate pathological complete response (pCR) in patients with metastatic uveal melanoma with resectable liver metastasis and absence of extrahepatic disease.
2. Which is the efficacy of tebentafusp used as a single agent to maintain disease control and delay relapse / progression.
3. Which is the safety of tebentafusp used as a single agent in metastatic uveal melanoma.

The main hypothesis is that neoadjuvant treatment with Tebentafusp could achieve ≥20% pathological complete response (pCR) in patients with metastatic uveal melanoma with resectable/potentially resectable liver metastasis and absence of extrahepatic disease. It is assumed that untreated patients would not present a pCR (response rate of ≤1%).

DETAILED DESCRIPTION:
1. RACIONAL Tebentafusp has demonstrated efficacy and safety and is indicated as monotherapy for the treatment of adult patients with human leukocyte antigen (HLA)-A*02:01-positive unresectable or metastatic uveal melanoma. The main hypothesis is that neoadjuvant treatment with Tebentafusp could achieve ≥20% pathological complete response (pCR) in patients with metastatic uveal melanoma with resectable or potentially resectable liver metastasis and absence of extrahepatic disease.
2. OBJECTIVES Primary Objective: to evaluate the ability of tebentafusp used as a single agent to generate pathological complete responses (pCR) in patients with metastatic uveal melanoma with resectable / potentially resectable liver metastases and absence of extrahepatic disease.

   Secondary objectives: to assess efficacy and safety of tebentafusp used as a single agent to maintain disease control and delay relapse / progression.

   Exploratory objectives:
   * Study mechanisms of resistance to tebentafusp.
   * Study correlation between pathological response and circulating tumor DNA (ctDNA) dynamics or circulating tumor cells (CTCs).
   * Evaluate dynamics in T-cell receptor (TCR) populations and peripheral lymphocytes memory cells in blood samples before/after Tebentafusp and in the prospective fresh samples from liver resections.
3. Primary Endpoint The primary endpoint for NEO-TB trial is the pathological complete response (pCR) rate, defined as no presence of residual disease assessed by biopsy or surgical resection at 7 months (+/-1 month) after the start of the scheduled treatment with tebentafusp.
4. Secondary Endpoints

   * Objective response rate (ORR) according to RECIST 1.1
   * Disease control rate (DCR) according to RECIST 1.1
   * Relapse-free survival (RFS) according to RECIST 1.1
   * Event-free survival (EFS)
   * Overall survival (OS)
   * Adverse events (AE)
   * Treatment-related AEs (TRAEs)
   * Molecular biomarkers determined from liver biopsies at baseline and fresh samples from liver resections in lesions with viable tumors and samples of peripheral blood.
5. Study Design

   NEO-TB is a non-randomized, single arm, multi-centre, phase II study of Tebentafusp monotherapy in subjects with resectable / potentially resectable disease within the liver and absence of extra-liver disease. The Neo-TB study is divided into 4 phases: Screening, Treatment, Surgery and Follow-up. After informed consent is obtained, subjects will enter the Treatment phase.

   All patients will undergo periodic tumor assessments by CT or MRI scan every 8 weeks ± 7 days from the start of study treatment and during the first 48 weeks of study. Tumor assessments will be performed every 12 weeks ± 7 days thereafter until relapse or patient withdrawal. After surgery, CT or MRI scans will be performed every 12 weeks ± 7 days thereafter, regardless of time after study inclusion. Further CT/MRI scans could be performed upon suspicion of disease relapse according to standard clinical practice and physician criteria. The study includes the collection of tumor and blood samples for the determination of exploratory endpoints
6. Study Population The trial will enroll 19 patients; male and female, ≥ 18 years, with ECOG PS 0-1 patients with metastatic uveal melanoma (HLA)-A*02:01 positive who have resectable or potentially resectable metastatic lesions only in the liver. Patients with extrahepatic disease are not eligible. Patients will have not received previously other anti-tumor treatments.
7. Study Treatment

   Patients will receive tebentafusp intravenously (IV) weekly for 6 months with liver directed imaging every 2 months to identify rapid progressors. Rapid progressors will discontinue tebentafusp and have surgical resection if considered feasible. After 6 months, patients with complete response (CR) according to RECIST will continue tebentafusp therapy (surgery might be an option if deem appropriate by local PI); while patients achieving partial response or stable disease will be evaluated for tumor resection and will enter into Surgery phase. Surgery will be conducted 7 months (+/- 1 month). If PD occurs earlier surgery can happen earlier. After surgery, patients without pCR or R0 surgery will maintain tebentafusp until disease relapse, unacceptable toxicity or patient withdrawal. Patients with pCR and R0 will continue tebentafusp therapy for 1 additional year or until disease relapse, unacceptable toxicity or patient withdrawal
8. Ethical Considerations Patients with metastatic uveal melanoma have limited therapeutic options. Clinical guidelines recommend considering clinical trials.

Tebentafusp is approved for use as monotherapy in patients with uveal melanoma whose tumors are positive for (HLA)-A*02:01. In the phase 3 clinical trial, tebentafusp showed a significant improvement in overall survival compared to other standard therapies and therefore it is considered the treatment of choice for patients with (HLA)-A*02:01 positive tumors.

NEO-TB aims to use tebentafusp in the pathology for which it is indicated, with the only modification of combining its administration with surgical resection in patients already or potentially candidates for surgery, aiming to evaluate the pathological response. The guidelines also allow this multimodal treatment strategy with tebentafusp and surgery, so the trial could in some way consider the proposed intervention as low impact. Patients will be closely monitored, following an adaptive strategy to allow surgery if necessary, avoiding delays that limit tumor resection. Tebentafusp is the standard therapy for these patients, so its administration in the context of this trial is not expected to increase the risks already described associated with this treatment. Given the mechanism of action of tebentafusp, an increase in its toxicity due to the combination with surgery is not expected. Immunotherapies in combination with surgery are used in the perioperative setting as neoadjuvant and adjuvant strategies in patients with cutaneous melanoma and are safe. However, there is no published data with patients treated with tebentafusp in this context.

Given the limited therapeutic options and the current evidence and rationale for the use of tebentafusp and surgery, the risk-benefit ratio of this trial is considered positive. The potential benefit outweighs the risks

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed metastatic uveal melanoma with Human leukocyte antigen-A*0201 positive determined by local assay.
2. Patients with histologically proven metastatic uveal melanoma in the liver with reectable or potentially resectable liver metastases evaluated by imaging in a multidisciplinary committee. Metastasis can be considered resectable by any of the following:

   1. Minor resection (i.e., less than a hemihepatectomy)
   2. Major resection (i.e., hemihepatectomy or extended hepatectomy)
   3. Bilobar resection (including atypical resection).
3. Must meet the following criteria related to prior treatment:

   1. No prior systemic therapy in the metastatic or advanced setting including chemotherapy, immunotherapy, or targeted therapy.
   2. No prior local, liver-directed therapy including chemotherapy, radiotherapy, radiofrequency ablation (RFA), or embolization.
   3. Prior neoadjuvant or adjuvant therapy is allowed provided it was administered in the curative setting in patients with localized disease.
4. Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written and signed informed consent.
5. Male or female patients age ≥ 18 years of age at the time of informed consent.
6. Eastern Cooperative Oncology Group Performance Status (ECOG-PS) 0-1
7. Adequate organ function as defined below (without transfusion):

   1. Hemoglobin ≥9.0 g/dL.
   2. Absolute neutrophil count (ANC) >1.5 x 109/L (> 1500 per mm3).
   3. Platelet count ≥ 100 x 109/L (>75,000 per mm3).
   4. Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with the Coordinating Investigator.
   5. Both AST and ALT must be < 5 x ULN.
   6. Creatinine clearance ⩾50 ml/min calculated by Cockcroft-Gault (Table 4) or another validated method.
   7. Potassium, magnesium, corrected calcium or phosphate abnormality of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) > grade 1.

Exclusion Criteria:

1. Presence of extrahepatic disease.
2. Patients with concomitant malignancy other than non-melanoma skin cancer, or superficial bladder cancer controlled with local treatment. Patients with prior malignancy must have been disease free for 5 years.
3. History of severe hypersensitivity reactions (eg, anaphylaxis) to other biologic drugs or monoclonal antibodies.
4. Clinically significant cardiac disease or impaired cardiac function, including any of the following:

   1. Clinically significant and/or uncontrolled heart disease such as congestive heart failure (New York Heart Association grade ≥ 2), uncontrolled hypertension, or clinically significant arrhythmia currently requiring medical treatment.
   2. QTcF > 470 msec on screening electrocardiogram (ECG) or congenital long QT syndrome.
   3. Acute myocardial infarction or unstable angina pectoris < 6 months prior to Screening.
5. History of adrenal insufficiency.
6. History of interstitial lung disease
7. History of pneumonitis that required corticosteroid treatment or current pneumonitis
8. History of colitis or inflammatory bowel disease.
9. Active infection requiring systemic antibiotic therapy. Patients requiring systemic antibiotics for infection must have completed therapy at least 1 week prior to the first dose of study drug.
10. Known history of human immunodeficiency virus (HIV) infection. Testing for HIV status is not necessary unless clinically indicated or if required by local regulations.
11. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection per institutional protocol. Testing for HBV or HCV status is not necessary unless clinically indicated.
12. Previous treatment with Tebentafusp.
13. Patients receiving systemic steroid therapy or any other immunosuppressive medication at any dose level. Local steroid therapies (eg, otic, ophthalmic, intra-articular or inhaled medications) are acceptable.
14. Major surgery within 2 weeks of the first dose of study drug (minimally invasive procedures such as bronchoscopy, tumor biopsy, insertion of a central venous access device, and insertion of a feeding tube are not considered major surgery and are not exclusionary).
15. Use of hematopoietic colony-stimulating growth factors (e.g., G-CSF, GMCSF, M-CSF) ≤ 2 weeks prior to the start of study drug. Patients must have completed therapy with hematopoietic colony-stimulating factor at least 2 weeks before the first dose of study drug is given. An erythroid-stimulating agent is allowed as long as it was initiated at least 2 weeks prior to the first dose of study treatment and the patient is not red blood cell transfusion dependent.
16. Hypersensitivity to the active substance of tebentafusp or to any of its excipients, including: Citric acid monohydrate (E330) Di-sodium hydrogen phosphate (E339) Mannitol (E421) Trehalose Polysorbate 20 (E432).
17. Patients whose circumstances will not permit study completion or adequate follow up.
18. Pregnant, likely to become pregnant, or lactating women (where pregnancy is defined as the state of a female after conception and until the termination of gestation).
19. Women of child-bearing potential who are sexually active with a non-sterilized male partner, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective contraception during study treatment, and must agree to continue using such precautions for 1 week after the final dose of investigational product. Highly effective methods of contraception are described in Appendix 5.
20. Male patients must be surgically sterile or use double barrier contraception methods from enrollment through treatment and for 1 week following administration of the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | Throughout the study period, at 7 months (+/- 1 month) from the start of treatment]
  Pathological complete response (pCR) rate, the primary efficacy endpoint: Defined as the rate of patients with metastatic uveal melanoma with resectable / potentially resectable liver metastasis and free of extrahepatic disease, who have no presence of residual disease assessed by biopsy or surgical resection at 7 months (+/- 1 month) after the start of the scheduled treatment with tebentafusp. pCR will be assessed locally on tumor samples from gross resection or biopsies obtained at 7 months (+/- 1 month) after the start of tebentafusp.

SECONDARY OUTCOMES:
Objective response rate (ORR) of neoadjuvant tebentafusp | Throughout the study period, at 6 months from the start of treatment
  Assessed by the investigator through imaging follow-up (CT scan/MRI) using RECIST 1.1 up to surgical intervention. This will be considered as the percentage/proportion of patients with complete response (CR) or partial response (PR) as their overall best response throughout the study period. Objective responses will be assessed locally by the investigator according to RECIST, version 1.1, and indicating the change in size of tumors as compared with baseline, before the first dose of study treatment.
Disease control rate (DCR) of neoadjuvant tebentafusp | Throughout the study period, at 6 months from the start of treatment
  Percentage/proportion of patients with complete response (CR) or partial response (PR), according to ORR definition for the trial, or maintained stable disease (SD) as their overall best response, assessed by imaging follow-up (CT scan/MRI) and RECIST 1.1 criteria. Stable disease should be maintained for at least 4 months to be considered as a DCR event. DCR will be assessed locally up to surgical intervention.
Relapse-free survival (RFS) at end of follow-up. | Throughout the study period, approximate average of 24 months since the start of treatment
  Defined as the time from first study dosing date to the date of relapse after surgery according to RECIST 1.1 (Appendix 3) or death due to any cause. Patients who do not have surgical resection will be not evaluable for RFS endpoint. The RFS will be estimated by the Kaplan-Meier method. Patients alive and free of events at the date of the analysis will be censored at their last known tumor assessment. Patients who start a new treatment line without progression will be censored on the date of first dose of the subsequent anticancer treatment. RFS will be displayed graphically where appropriate.
  RFS will be calculated as median / mean (95% CI) and for different timepoints:
  * Proportion of patients without relapse at the end of follow-up.
  * Proportion of patients relapse-free at 6-months, 12-months and as deemed opportune by the time of the analysis
  The Cox proportional hazards model will be fitted to compute the hazard ratios on potential stratified groups if applicable.
Relapse-free survival (RFS) at at 6-months | Throughout the study period, at 6 months from the start of treatment
  Defined as the time from first study dosing date to the date of relapse after surgery according to RECIST 1.1 (Appendix 3) or death due to any cause. Patients who do not have surgical resection will be not evaluable for RFS endpoint. The RFS will be estimated by the Kaplan-Meier method. Patients alive and free of events at the date of the analysis will be censored at their last known tumor assessment. Patients who start a new treatment line without progression will be censored on the date of first dose of the subsequent anticancer treatment. RFS will be displayed graphically where appropriate.
  RFS will be calculated as median / mean (95% CI) and for different timepoints:
  * Proportion of patients without relapse at the end of follow-up.
  * Proportion of patients relapse-free at 6-months, 12-months and as deemed opportune by the time of the analysis
  The Cox proportional hazards model will be fitted to compute the hazard ratios on potential stratified groups if applicable.
Relapse-free survival (RFS) at 12 months | Throughout the study period, at 12 months from the start of treatment
  Defined as the time from first study dosing date to the date of relapse after surgery according to RECIST 1.1 (Appendix 3) or death due to any cause. Patients who do not have surgical resection will be not evaluable for RFS endpoint. The RFS will be estimated by the Kaplan-Meier method. Patients alive and free of events at the date of the analysis will be censored at their last known tumor assessment. Patients who start a new treatment line without progression will be censored on the date of first dose of the subsequent anticancer treatment. RFS will be displayed graphically where appropriate.
  RFS will be calculated as median / mean (95% CI) and for different timepoints:
  Proportion of patients relapse-free at 6-months, 12-months and as deemed opportune by the time of the analysis
  The Cox proportional hazards model will be fitted to compute the hazard ratios on potential stratified groups if applicable.
Overall survival (OS) | Throughout the study period, at 12 months from the start of treatment
  Defined as the time elapsed from the first dose of study treatment until death from any cause. Patients alive and free of events at the date of the analysis will be censored at their last known contact. OS will be summarized using the Kaplan-Meier method and displayed graphically where appropriate. The Cox proportional hazards model will be fitted to compute the hazard ratios on potential stratified groups if applicable. OS will be calculated as median / mean (95% CI) and OS rate for different timepoints deemed appropriate at the time of the analysis (i.e.1-year OS rate) will also be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Maria Piulats, M.D., Ph.D., Study Chair — Institut Catala d'Oncologia (ICO) Hospitalet
Locations (4):
- Charité - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany
- Spain (3):
  - Institut Catala d'Oncologia (ICO) Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital La Paz, Madrid, Madrid
  - Consorcio Hospital General Universitario de Valencia, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No